CLINICAL TRIAL: NCT06012214
Title: Robot-assisted Versus Conventional Minimally Invasive Esophagectomy for Locally Advanced Esophageal Squamous Cell Carcinoma After Neoadjuvant Therapy: a Prospective Randomized Controlled Trial
Brief Title: RAE Versus MIE in Patients With Esophageal Cancer After Neoadjuvant Therapy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Zhigang Li, Prof., Shanghai Chest Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RAMIE-2
Record Dates: First submitted 2023-06-15; First posted 2023-08-25 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Surgical Procedure, Unspecified

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robot-assisted minimally invasive esophagectomy (Experimental): Participants will received neoadjuvant therapy followed by robot-assisted minimally invasive esophagectomy within 8 weeks.
  Interventions: Procedure: ROBOTIC-ASSISTED ESOPHAGECTOMY
- Thoraco-laparoscopic minimally invasive esophagectomy (Placebo Comparator): Participants will received neoadjuvant therapy followed by thoraco-laparoscopic minimally invasive esophagectomy within 8 weeks.
  Interventions: Procedure: ROBOTIC-ASSISTED ESOPHAGECTOMY

INTERVENTIONS:
Procedure: ROBOTIC-ASSISTED ESOPHAGECTOMY — Comparison between robotic and conventional minimally invasive esophagectomy

SUMMARY:
This is a prospectively randomized controlled trial to compare RAMIE and MIE in the treatment for locally advanced ESCC after neoadjuvant therapy. According to previous studies, long-term survival after RAMIE seemed to be at least comparable to MIE or open esophagectomy. Therefore, the RAMIE-2 study was designed as a non-inferiority trial, which was based on the hypothesis that the 5-year overall survival of patients who received RAMIE is uncompromised to MIE. To achieve the primary endpoint, 260 cases will be recruited in our hospital. Based on the volume of esophagectomy (1000 cases/year) and the proportion of patients with neoadjuvant therapy (50%) in our institution, approximately 10 patients will be enrolled for each group per month for this trial. The study will be performed in accordance with the principles of the Declaration of Helsinki and Good Clinical Practice Guidelines. Written informed consent will be obtained from each participant. The flow chart of this trial is also presented.

DETAILED DESCRIPTION:
Neoadjuvant therapy followed by radical resection is the recommended treatment for locally advanced esophageal cancer, which could achieve a better R0 resection and overall survival. With the development of multidisciplinary treatment of esophageal cancer, especially the emerging concept of "watch and wait", surgery may only be a new era of salvage treatment for patients with poor response to neoadjuvant or recurrence after definitive treatment in the future. At that time, the technical advantage of RAMIE should be even more valuable. Early results of the RAMIE trial (conducted by our group)15, has demonstrated that RAMIE can achieve shorter operative time as well as better lymph node dissection in patients who received neoadjuvant therapy, compared to conventional MIE. In addition, this benefit was more obviously observed in lymph nodes along the bilateral recurrent laryngeal nerves, which were considered as the most challenging steps.

Therefore, we put forward a hypothesis: whether the robot's superior human-surgical interface is beneficial to achieve better surgical and oncological results in patients with locally advanced ESCC after neoadjuvant therapy. Based on the results of RAMIE trial, the present RAMIE-2 study is trying to answer such a question.

ELIGIBILITY:
Inclusion Criteria:

1. Age ranges from 18 to 75 years;
2. European Clinical Oncology Group Performance Status (ECOG PS) 0-2;
3. Histological subtype of esophageal squamous cell carcinoma;
4. Primary tumors are located at the intrathoracic esophagus;
5. Pre-treatment stage as cT1b-4aN1-3M0, cT3N0M0 (AJCC/UICC 8th Edition);
6. With neoadjuvant chemoradiotherapy, chemotherapy and immunotherapy;
7. Without any anticancer therapy for other malignant diseases;
8. Written informed consent.

Exclusion Criteria:

1. Cervical esophageal cancer and carcinoma of gastro-esophageal junction;
2. Patients with unresectable or metastatic esophageal cancer;
3. Histological subtype of esophageal non-squamous cell carcinoma;
4. History of previous thoracic surgery;
5. Patients with other malignant tumor (previous or current);
6. Participation in another clinical trial during this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
overall survival | up to 5 years
  defined as the time from the date of surgery to the day of death or to the last follow-up.

SECONDARY OUTCOMES:
disease-free survival | up to 5 year
  defined as the time from the date of surgery to the day of tumor recurrence, tumor progression or death assessed up to 5 years
oncologic results | 4 weeks
  number of lymph nodes dissection, R0 resection rate

CONTACTS AND LOCATIONS:
Overall Officials: Zhigang Li, Dr., Principal Investigator — Shanghai Chest Hospital
Locations (1):
- Shanghai Chest Hospital, Shanghai Jiao Tong University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No